CLINICAL TRIAL: NCT06467370
Title: CONFIDENCE: A Prospective Observational Study With Acute Treatment of Rimegepant ODT on Consistency, Satisfaction and Tolerability of Treatment in the Real World
Brief Title: A Real-world, Prospective Observational Study of Rimegepant ODT for the Acute Treatment of Migraine Attacks in Adults.
Acronym: CONFIDENCE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Aptar Digital Health (Industry)
Responsible Party: Sponsor
Other Study IDs: C4951072; AUDACITY (Other: Alias Study Number)
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: rimegepant; acute migraine treatment; real-world setting
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biosamples will be collected in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at characterizing the effectiveness of rimegepant as an acute migraine treatment in a real world setting on two aspects:

* Consistency of response to rimegepant across multiple attacks
* Effectiveness of rimegepant in users taking concomitant migraine preventive medications, namely monoclonal antibodies targeting CGRP and onabotulinumtoxinA

DETAILED DESCRIPTION:
This study will be conducted in a real-world setting in the US using a bespoke interface contained in the Migraine Buddy mobile application. Participants who report using rimegepant for the acute treatment of migraine will be recruited and will be asked to complete a series of questionnaires during the screening and study period. Patient reported outcome measures will be collected at study enrollment, daily during the 28-day observation period, and at the end of the study period.

Research Questions:

1. In adult patients currently receiving a prescription for rimegepant for the acute treatment of migraine, what is the population-level consistency of rimegepant response for pain reduction, meaningful pain relief, performance in daily activities, and return to normal function across multiple attacks in a real-world setting, regardless of prophylactic background?
2. What is the satisfaction level of patients receiving rimegepant on background migraine prophylaxis (specifically, anti-CGRP mAbs or onabotulinumtoxinA (Botox)?
3. What is the efficacy, safety, and tolerability of rimegepant for the acute treatment of migraine, when taken in combination with preventive medications that act on the same pathway?

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with migraine ≥18 years old
* Having received a prescription for rimegepant for acute treatment
* Experienced between 3 and 14 Headache days in the last 30 days
* Planning to use rimegepant for attacks happening during the next 30 days

Exclusion Criteria:

* Report currently using rimegepant as preventive
* Report currently using concomitantly onabotulinumtoxin and any of the mAbs
* Currently participating in a Migraine-related clinical trial
* Reports a diagnosis from a doctor or other health professional of cluster headache, post-traumatic headache, new daily persistent headache, or hemicrania continua

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 4 subpopulations in this study:
  1. participants using rimegepant and no prophylactic
  2. participants using rimegepant with background prophylaxis of OMPM
  3. participants using rimegepant with background prophylaxis of mAbs
  4. participants using rimegepant with background prophylaxis of Botox.
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Satisfaction with prescribed medication | Day 30
  Satisfaction with prescribed medication (rimegepant-treated attacks) as measured by 5 questions with a 7-point rating scale; Distribution analysis and Responder Yes/No. Responder definition: Extremely Satisfied, Satisfied, Slightly Satisfied."
Population level consistency | Day 30
  Population level consistency will be determined utilizing the daily diary item 'meaningful pain relief' when rimegepant is used to acutely treat a migraine attack. Those who report meaningful pain relief at <1 or 1-2 hours after taking rimegepant will be considered a 'responder'. Those who report meaningful pain relief >2 hours or those who did not achieve meaningful relief/used another acute treatment since taking rimegepant will be considered 'delayed responder' or 'non-responder,' respectively. Population level consistency will be evaluated as the proportion of responders for each attack treated with rimegepant.
Assessments of meaningful clinical effect | Day 30
  Assessments of meaningful clinical effect will be measured by the rates in achieving meaningful pain relief at other timepoints, rates of improvement of migraine severity and functional disability, satisfaction with treatment and rates of acute treatment optimization. Responder definition: Improvement in functional disability 2 hours after taking rimegepant vs at time of intake (reduction by at least 1 category:e.g., from severely impaired to moderately impaired, from moderately impaired to mildly impaired, from mildly impaired to no disability).
meaningful improvement in functioning | Day 30
  Experience of "meaningful improvement in functioning" between 1 and 4 hours after intake.

SECONDARY OUTCOMES:
Effectiveness of rimegepant in users taking concomitant migraine preventive medications | Day 30
  Percentage of Participants Achieving Meaningful Pain Relief Meaningful relief occurs when the level of headache pain has been reduced to a degree that is meaningful to the participant; this can, but does not necessarily, occur prior to pain freedom. Participants will provide responses for rimegepant-treated migraine attacks about the time to achieve meaningful relief of headache pain. This will result in a binary responder definition coded as "yes" for those achieving meaningful pain relief or "no" for those not satisfying that definition.
  Percentage of Participants Who Experience Meaningful improvement in functioning Participants will also rate the ability to perform daily activities at the point when rimegepant was taken using the Functional Disability Scale. This will result in a binary responder definition coded as "yes" for those achieving return to normal function or "no" for those not satisfying that definition.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951072